CLINICAL TRIAL: NCT05079087
Title: Pericapsular Nerve Group Block for Positional Pain and Postoperative Analgesia
Brief Title: Pericapsular Nerve Group Block for Positional Pain and Postoperative Analgesia in Hip Fractures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Azienda Sanitaria dell'Alto Adige (Other)
Responsible Party: Principal Investigator, Paolo Seraglio, Principal Investigator, Azienda Sanitaria dell'Alto Adige
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 01
Record Dates: First submitted 2021-03-04; First posted 2021-10-15 (Actual); Last update posted 2021-10-15 (Actual); Status verified 2021-10

CONDITIONS: Pertrochanteric Fracture; Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PENG BLOCK arm (Experimental): The first arm will consist of patients that undergo PENG block administering a mixture of Ropivacaine 0.5% + Dexamethasone 4 mg in a volume of 20 ml before performing the spinal anaesthesia.
  Interventions: Procedure: Pericapsular nerve group blockade
- Ketamine- Midazolam arm (Active Comparator): The second arm consist in Patients that will undergo sedation and analgesic treatment with Ketamine and Midazolam titrated to the best Verbal Rating Score without respiratory and cardiovascular depressant effect.
  Interventions: Drug: Midazolam Ketamine arm

INTERVENTIONS:
Procedure: Pericapsular nerve group blockade — The PENG-block will be administered under ultrasound (US) guidance with a low frequency curvilinear probe. The probe will be placed parallel to the inguinal crease at the level of the anterior superior iliac spine. Scanning will be done with gradual caudal movement of the probe. After the anterior inferior iliac spine (AIIS) is visible, the probe will be turned slightly medial until the hyperechoic continuous shadow of the superior pubic ramus is visible. The Psoas muscle with its prominent tendon will be identified just above the pubic ramus. The target is the plane between the 2 structures. While aligning the pubic ramus in the center of the image and targeting the pubic ramus just medial to the AIIS, a 22 Go 10 cm needle will be introduced and 20 ml of anesthetic solution administered.
  Other Names: PENG block
  Arms: PENG BLOCK arm
Drug: Midazolam Ketamine arm — Patients in the second group will undergo sedation and analgesic treatment with Ketamine and Midazolam titrated to the best Verbal Rating Score without respiratory and cardiovascular depressant effect.
  Other Names: Analgosedation treatment
  Arms: Ketamine- Midazolam arm

SUMMARY:
The aims of this study are:

* Evaluate the effectiveness of the pericapsulare blockade of the femoral nerve, the accessory obturator nerve and the obturator nerve in patients with pertrochanteric fractures of the femur, during the pre-operative period for patient positioning manoeuvres (sitting position for performing spinal anaesthesia, mobilisation on the operating bed, etc.);
* Evaluate the consumption of opioids or hypnotics in the perioperative period, which are more responsible for the incidence of delirium in the elderly patient;
* Evaluate the duration and quality of postoperative analgesia and well-being.

DETAILED DESCRIPTION:
Pertrochanteric femoral fracture is a frequent orthopaedic emergency in the elderly and is associated with significant morbidity and mortality. Surgical reduction and subsequent fixation is the definitive therapy for most patients. Recent clinical studies show that early treatment within the first 48 hours significantly reduced mortality and major complication (pulmonary embolism, sepsis, cardiac events, renal and respiratory failure). Even though, data regarding the anaesthesiology method best suited for this intervention are somewhat controversialthe Italian Society for Anaesthesiology, Analgesia Reanimation and intensive care recommends spinal anaesthesia as the standard procedure. In addition, the Association of Anaesthetists of Great Britain and Ireland recommend this approach.

Patient mobilisation for the administration of spinal anaesthesia as well as post-operative care require effective perioperative pain management. In current practice, this is achieved by the administration of systemic analgosedative treatment. Ideally, the use of opioids or ketamine should be minimized since their side effects are major morbidity factors. Peripheral nerve blocked can be an efficient to foster pre- and postoperative analgesia and therefore minimize the need for opioids.

Currently, the psoas compartment block is considered to be the most reliable peripheral nerve block for analgesia in pertrochanteric femoral fractures, although it is technically rather difficult to perform and could be associated with serious side effects. Alternative approaches, such as the femoral nerve block, the Iata band block or the 3-in-1 block often do not possess a sufficient reliable analgesic effect in this kind of injury. Thus so far, peripheral nerve blocks are not routinely applied in clinical practice in most cases.

The anterior capsule of the hip joint is the most innervated area of the entire joint.

The nerves involved are:

* The obturatorial nerve
* The accessory nerve of the obturator
* The femoral nerve Adequate anaesthesia for pertrochanteric femoral facture requires the blockage of all three nerves. In 2018, Gíron-Arango et al., developed a novel ultrasound guided approach for the blockade these nerves, the Pericapsular nerve group (PENG) block. The investigators consider this peripheral nerve block a potentially beneficial technique to implement in the treatment of per trochanteric femur fracture patients.

Patients with a pertochanteric femoral fracture admitted to the orthopaedics department for surgical treatment will be asked whether they are willing to participate to the study. After transfer of the patient to Anaesthesiology, before performing any additional analgesic measures, the NRS at rest and on the movement of the affected limb (extension of 20°) will be evaluated. The 4AT test for the assessment of delirium will be performed to obtain a baseline value. The participants will be randomly assigned to two groups. Due to the fact that these patients need swift treatment for their injury, our randomisation is based on alternating assignments to the two groups based on the time patients sign their informed consent for study participation. The investigators have no indication that this randomisation procedure could lead to a bias. The first group will consist of patients that undergo PENG block administering a mixture of Ropivacaine 0.5% + Dexamethasone 4 mg in a volume of 20 ml before performing the spinal anaesthesia. There is one report indicating that a 1:1 mixture of ropivacaine 0.75% with 4mg/mL dexamethasone could pose a risk due to crystal formation. However, in our clinical practice, where the investigators mix 0.5% in a 1:20 ratio, thus producing an injection containing 30-times less dexamethasone, the investigators did never experience problems with crystallisation. This is extensively backed by literature. In any case, the patients will be informed about the off-label nature of perineural dexamethasone during the anaesthesiologic visit.

The PENG-block will be administered under ultrasound (US) guidance with a low frequency curvilinear probe. The probe will be placed parallel to the inguinal crease at the level of the anterior superior iliac spine. Scanning will be done with gradual caudal movement of the probe. After the anterior inferior iliac spine (AIIS) is visible, the probe will be turned slightly medial until the hyperechoic continuous shadow of the superior pubic ramus is visible. The Psoas muscle with its prominent tendon will be identified just above the pubic ramus. The target is the plane between the 2 structures. While aligning the pubic ramus in the center of the image and targeting the pubic ramus just medial to the AIIS, a 22 Go 10 cm needle will be introduced and 20 ml of anesthetic solution administered. The participants are informed about the specifics of the PENG blocks and the risks (which are minor) during the anesthesiologic visit.

Patients in the second group will undergo sedation and analgesic treatment with Ketamine and Midazolam titrated to the best Verbal Rating Score without respiratory and cardiovascular depressant effect. 30 minutes after the PENG block or the drug treatment, immediately before mobilization for the spinal anaesthesia, the assessment of NRS at rest and on movement of the affected limb (extension of 20°) will be repeated.

Spinal anaesthesia will be performed using 2.5mL isobaric bupivacaine 0.5% applying state of the art care.

After surgical intervention in postoperative care, patients do not receive fix systemic analgesia as post-operative pain should be covered by the PENG block. However, in the post-operative are they will receive Paracetamol, Metamizole and Buprenorphine if necessary. Once they are transferred to the orthopaedics department, patients analgesia will be managed according to the orthopaedics department standardized protocols. In any case, post-operative opiate consumption will be recorded. To assess post-operative pain management performance in the two groups, the NRS at rest and on movement of the affected limb (extension of 20°) will be evaluated 18 hours after the PENG block. In order to avoid too much discomfort for the patients and to not induce unnecessary inflammation in the surgical area, the investigators refrain of doing too many measurements. The investigators expect that the the 18 hours measurement together with the evaluation of post-operative opiate use will give us a clear image of post-operative pain control. Also, 18 hours after, the 4AT test will be performed to quantify symptoms of delirium. Furthermore, the occurrence of PONV and patient satisfaction on a VAS-Scale will be evaluated.

The primary endpoint is the NRS variations during movement of the affected limp (extension of 20°) before and 30 minutes as well as 18 hours after performing the PENG block or analgosedation. Secondary endpoints are occurrence of delirium quantified by the 4AT test, if and who much and which rescue opiate was used, occurrence of PONV and patient satisfaction expressed on a VAS-Scale.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a peritrocanteric femur fracture admitted to the orthopaedic ward

Exclusion Criteria:

* Patient refusal
* Lack of informed consent
* Pathological skin alterations
* Intertrigo at the puncture site level.
* Allergy to any of the drugs
* Coagulopathy
* Sepsis
* Use of direct oral anticoagulatns (DOACs)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-04-01 (Estimated); Study Completion 2022-11-01 (Estimated)

PRIMARY OUTCOMES:
Change of the numerical rating scale for pain (NRS) during movement of the affected limb (extension of 20°) 30 minutes after the PENG block | Change in NRS pre and 18 hours post performing the PENG block

SECONDARY OUTCOMES:
Delirium | Changne in score of the 4 AT rapid clinical test pre and 18 hours post performing block
  Change in score of the rapid assessment test for delirium screening
Rescue opiate use | During the first 24 hours after discharge from the recovery room
  Evaluate the use of opioids in the postoperative period.
PONV | During the first 24 hours after discharge from the recovery room
  Record the occurrence of nausea or vomiting
Questionnaire on patient satisfaction | From the beginning of the surgical procedure until 24 hours after discharge from the recovery room
  Evaluate subjective patient satisfaction

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda sanitaria Allo Adige ospedale di Merano, Meran, Bolzano, Italy

IPD SHARING:
Plan to Share IPD: Undecided